CLINICAL TRIAL: NCT03851952
Title: Re-Establishing Flow Via Drug Coated Balloon for the Treatment of Urethral Stricture Disease - Registry Study
Acronym: ROBUST IV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company Decision
Sponsor: Urotronic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR1117
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Urethral Stricture; Urethral Stricture, Anterior; Lower Urinary Tract Symptoms; Anterior Urethral Stricture
MeSH Terms: conditions — Urethral Stricture; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Optilume DCB (Other): Optilume Drug Coated Balloon (DCB) treatment for the treatment of urethral stricture as approved for use in Canada
  Interventions: Device: Optilume Drug Coated Balloon

INTERVENTIONS:
Device: Optilume Drug Coated Balloon — The Optilume Drug Coated Balloon (DCB) is a guidewire compatible catheter with a tapered atraumatic tip. The distal end of the catheter has an inflatable balloon coated with a proprietary coating containing the drug paclitaxel that facilitates the drug's transfer to the urethral wall upon inflation.

SUMMARY:
The ROBUST IV study is designed to collect and better understand "real-world" outcomes for men undergoing urethral dilation using the Optilume Drug Coated Balloon (DCB) for treatment of urethral stricture.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥ 18 years old
2. Visual confirmation of stricture via cystoscopy or retrograde urethrogram
3. Single lesion bulbar urethral stricture, less than or equal to 3.0 cm
4. Significant symptoms of stricture such as frequency of urination, dysuria, urgency, hematuria, slow flow, feeling of incomplete emptying, recurrent urinary tract infections (UTIs).
5. IPSS score of 13 or higher
6. Lumen diameter <12F by urethrogram
7. Able to complete validated questionnaire independently
8. Qmax <15 ml/sec
9. Guidewire must be able to cross the lesion

Exclusion Criteria:

1. Strictures greater than 3.0 cm long
2. Subjects with greater than 1 stricture.
3. Sensitivity to paclitaxel or on medication that may have negative interaction with paclitaxel
4. Previous urethroplasty within the anterior urethra
5. Stricture due to bacterial urethritis
6. Stricture due to untreated gonorrhea
7. Stricture due to Lichen Sclerosus, or balanitis xerotica obliterans (BXO)
8. Stricture dilated or incised within the last 3 months (apart from subjects on self-catheterization)
9. Presence of local adverse factors (e.g. abnormal prostate, urethral false passage or fistula) making catheterization difficult
10. Presence of signs of obstructive voiding symptoms not directly attributable to the stricture at the discretion of the physician
11. Diagnosis of untreated and unresolved severe BPH or bladder neck contracture (BNC), at the discretion of the physician
12. Prior diagnosis of overactive bladder (OAB)
13. Diagnosis of severe stress urinary incontinence (SUI), at the discretion of the physician
14. Previous radical prostatectomy that resulted in either unresolved bladder neck contracture (BNC) and/or unresolved incontinence
15. Previous pelvic radiation
16. Diagnosis of kidney, bladder, urethral or ureteral stones in the last 6 weeks or active stone passage in the past 6 weeks
17. Diagnosed with chronic renal failure, at the discretion of the physician
18. A dependence on Botox (onabotulinumtoxinA) in the urinary system
19. Presence of a penile implant, artificial urinary sphincter, or stent(s) in the urethra or prostate
20. Known neurogenic bladder, sphincter abnormalities, or poor detrusor muscle function
21. Previous hypospadias repair
22. Diagnosis within the last 5 years of carcinoma of the bladder or prostate or suspicion of prostate cancer (e.g. abnormal DRE or high PSA) at the discretion of the physician
23. Any cognitive or psychiatric condition that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affect the ability to complete the study quality of life questionnaires
24. Unwilling to use protected sex for ≥30 days post treatment
25. Unwilling to abstain or use protected sex for 90 days post treatment if sexual partner is of child bearing potential.
26. Inability to provide legally effective Informed Consent Form (ICF) and/or comply with all the required follow-up requirements
27. Active infection in the urinary system
28. History of diabetes not controlled with a hemoglobin A1-C >7.0%
29. Diagnosed or suspected primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function, sphincter function or poor detrusor muscle function.
30. Visible hematuria with subject urine sample without known contributing factor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-31 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Stricture Recurrence Rate | 12 months
  Stricture Free Rate
Rate of Serious Adverse Events | 3 months
  Major Device or Procedure Related Serious Adverse Events

SECONDARY OUTCOMES:
Change in Uroflow | 3 and 12 months
  Change in Qmax (peak flow rate)
Change in the International Prostate Symptom Score Questionnaire (IPSS) | 3 and 12 months
  IPSS Percent Responder (50% improvement in IPSS score or IPSS score of 11 or lower)
Change in the EQ-5D Quality of Life Questionnaire | 3 and 12 months
  Change in the EQ-5D at 3 and 12 months post-procedure compared to baseline. Subscales of mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale of 1 (no problem) to 5 (extreme problems)
Change in the International Index of Erectile Function Questionnaire (IIEF) | 3 and 12 months
  Change in the IIEF at 3 and 12 months post-procedure compared to baseline on a scale of 5 (severe erectile dysfunction) to 25 (no erectile dysfunction)
Change in the Male Sexual Health Questionnaire (MSHQ-EjD) | 3 and 12 months
  Change in the MSHQ-EjD at 3 and 12 months post-procedure compared to baseline. Subscales of ejaculatory function from 1 (more ejaculatory dysfunction) to 15 (less ejaculation dysfunction) and bother from 0 (no bother with ejaculation) to 5 (greater bother with ejaculation)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Kodama, MD, Principal Investigator — Sunnybrook Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No